CLINICAL TRIAL: NCT00287404
Title: A Comparison of NMR and Chemical Lipid Analysis in the Fasting and Postprandial State in Patients With Type 2 Diabetes
Brief Title: Measuring Cholesterol in the Fasting and Postmeal State in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of North Carolina (Other)
Collaborators: LipoScience, Inc. (Industry)
Organization: University of North Carolina, Chapel Hill (Other)
Other Study IDs: GCRC-2395; GCRC-2395
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; hyperlipidemia; dyslipidemia; fasting lipids; postprandial lipids; Non-HDL cholesterol; NMR lipoanalysis; ATP III guidelines
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperlipidemias; Dyslipidemias

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Many patients with type 2 diabetes have difficulty attaining cholesterol goals, partly due to the recommendations for fasting measurements that may not be practical in the typical clinical setting. Focus toward therapy is shifting toward non-fasting assessments but little is known about the usefulness of this approach in diabetes, where postmeal cholesterol levels are more abnormal. This is an observational study examining fasting and postmeal lipids (cholesterol) in patients with type 2 diabetes using standard means and NMR.

DETAILED DESCRIPTION:
Current treatment guidelines for dyslipidemia focus on fasting lipid panels, specifically LDL cholesterol (LDL) but compliance has been shown to be poor. Therefore, focus has shifted to non-fasting measurements. However, there has been limited data in patients with type 2 diabetes and further study is needed to illuminate the lipid changes that occur in the non-fasting state. This observational study examines fasting and postprandial lipids in patients with type 2 diabetes using standard chemical analysis and NMR. For comparison, lipid panels will be obtained at baseline and 3 hours following a standard meal in 30 patients with type 2 diabetes. These measurements will then be analyzed based on current ATP III guidelines. We will investigate the degree to which the postprandial assessments agree with the fasting assessments and the agreement between LDL and the two alternative measures --- non-HDL and NMR-LDL.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75
* male or female
* Type 2 diabetes
* Hemoglobin A1C less than 9 at last measurement (within 3 months)

Exclusion Criteria:

* Pregnancy
* Non-English speaking.
* Inability to fast for 12 hours
* Hypoglycemia requiring assistance in the previous 6 months
* Unwilling to consume the standardized meal

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-10; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: John Buse, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Diabetes Care Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Bottorff MB. Underidentification and undertreatment issues. J Manag Care Pharm. 2003 Jan-Feb;9(1 Suppl):6-8. doi: 10.18553/jmcp.2003.9.s1.6. PMID 14613352
- [Background] Craig SR, Amin RV, Russell DW, Paradise NF. Blood cholesterol screening influence of fasting state on cholesterol results and management decisions. J Gen Intern Med. 2000 Jun;15(6):395-9. doi: 10.1046/j.1525-1497.2000.03509.x. PMID 10886474
- [Background] Bittner V. Non-high-density lipoprotein cholesterol: an alternate target for lipid-lowering therapy. Prev Cardiol. 2004 Summer;7(3):122-6; quiz 129-30. doi: 10.1111/j.1520-037x.2004.3094.x. PMID 15249764
- [Background] Iovine C, Vaccaro O, Gentile A, Romano G, Pisanti F, Riccardi G, Rivellese AA. Post-prandial triglyceride profile in a population-based sample of Type 2 diabetic patients. Diabetologia. 2004 Jan;47(1):19-22. doi: 10.1007/s00125-003-1269-3. Epub 2003 Nov 26. PMID 14647893
- [Background] Teno S, Uto Y, Nagashima H, Endoh Y, Iwamoto Y, Omori Y, Takizawa T. Association of postprandial hypertriglyceridemia and carotid intima-media thickness in patients with type 2 diabetes. Diabetes Care. 2000 Sep;23(9):1401-6. doi: 10.2337/diacare.23.9.1401. PMID 10977041
- [Background] Weiss R, Harder M, Rowe J. The relationship between nonfasting and fasting lipid measurements in patients with or without type 2 diabetes mellitus receiving treatment with 3-hydroxy-3-methylglutaryl-coenzyme A reductase inhibitors. Clin Ther. 2003 May;25(5):1490-7. doi: 10.1016/s0149-2918(03)80134-0. PMID 12867223
- [Background] Garvey WT, Kwon S, Zheng D, Shaughnessy S, Wallace P, Hutto A, Pugh K, Jenkins AJ, Klein RL, Liao Y. Effects of insulin resistance and type 2 diabetes on lipoprotein subclass particle size and concentration determined by nuclear magnetic resonance. Diabetes. 2003 Feb;52(2):453-62. doi: 10.2337/diabetes.52.2.453. PMID 12540621
- [Background] Tsai MY, Georgopoulos A, Otvos JD, Ordovas JM, Hanson NQ, Peacock JM, Arnett DK. Comparison of ultracentrifugation and nuclear magnetic resonance spectroscopy in the quantification of triglyceride-rich lipoproteins after an oral fat load. Clin Chem. 2004 Jul;50(7):1201-4. doi: 10.1373/clinchem.2004.032938. Epub 2004 May 13. PMID 15142979
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Derived] Dungan KM, Guster T, DeWalt DA, Buse JB. A comparison of lipid and lipoprotein measurements in the fasting and nonfasting states in patients with type 2 diabetes. Curr Med Res Opin. 2007 Nov;23(11):2689-95. doi: 10.1185/030079907x233304. PMID 17892636